CLINICAL TRIAL: NCT04803981
Title: Infancy to Toddlerhood: Early Nutrition & Tolerance (INTENT)
Acronym: INTENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Before Brands, Inc (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SF-003
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Diet Diversity; Infant Nutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard diet with daily SpoonfulONE (Experimental): Participants will receive one serving of SO (one of three possible forms of SO: mix-ins, puffs, or crackers) daily in addition to a standard diet. The SO form fed on a given day will be at the discretion of the parent/guardian.
  Interventions: Other: SpoonfulONE
- Standard diet (No Intervention): Participants will feed on a standard diet only, with no intervention, and complete questionnaires

INTERVENTIONS:
Other: SpoonfulONE — SpoonfulONE is a line of nutritional food products designed to help improve diet diversity starting in early infancy. SpoonfulONE covers a wide range of food proteins. Each product contains 30 mg of peanuts, milk, shellfish (shrimp), tree nuts (almond, cashew, hazelnut, pecan, pistachio, and walnut), egg, fish (cod and salmon), grains (wheat and oat), soy, and sesame.
  Arms: Standard diet with daily SpoonfulONE

SUMMARY:
This is a randomized, controlled, open-label, pragmatic, direct-to-participant trial designed for infants. The study will be conducted using a mobile application platform to engage parents with healthy infants and parents with infants with eczema in introducing complementary feeding in line with new feeding guidelines for diet diversity, gather parental experiences of feeding, support early introduction of different food proteins and support feeding of SpoonfulONE.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 4-6 months of age at time of consent
2. Provision of signed and dated informed consent form parent/guardian(s)
3. Parent/guardian(s) stated willingness to introduce within 12 months and feed the participant 5 common foods, including peanuts, cashew, egg, sesame, and cod
4. In good general health as evidenced by medical history reported by the parent/guardian(s)
5. No known allergy to any of the ingredients in the study intervention (SO), their components, or excipients

Exclusion Criteria:

1. Known physician confirmed allergies to any of the ingredients in SO at the time of consent
2. Gastroesophageal reflux disease (GERD) diagnosed by a physician and requiring treatment (i.e., pharmacological and/or non-pharmacological treatments such as a wedge)
3. Participant or parent/guardian unsuitable for the study, at the discretion of the investigator
4. Sibling in the home is already enrolled in the study

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of foods tolerated by participants, measured through a feeding questionnaire, of 5 common foods (peanut, egg, cashew, cod, and sesame) | 12 months
  Proportion of foods tolerated by participants, measured through a feeding questionnaire, of 5 common foods (peanut, egg, cashew, cod, and sesame)

SECONDARY OUTCOMES:
Parent/guardian comfort level of introducing food proteins into the participant's diet, Likert score | Baseline
  Parent/guardian comfort level of introducing food proteins into the participant's diet, Likert score
Diet diversity, score | 12 months
  Diet diversity score measured through regular questionnaires where participants will indicate which foods they are eating
Mean age of participants when first introduced to various food groups, measured through a questionnaire | 12 months
  Mean age of participants when first introduced to various food groups, measured through a questionnaire
Convenience, score through a questionnaire | 12 months
  Convenience of using daily SpoonfulONE, measured through a questionnaire
Proportion of participants compliant to daily feeding protocols, measured through a questionnaire | 12 months
  Proportion of participants compliant to daily feeding protocols, measured through a questionnaire
Proportion of foods tolerated by participants, measured through a feeding questionnaire, of 9 common food groups | 12 months and 18 months
  Proportion of foods tolerated by participants, measured through a feeding questionnaire, of 9 common food groups
Proportion of participants on SpoonfulONE compared to the proportion of participants on the non-intervention arm who tolerated each individual food groups of the 9 selected food groups, measured through a questionnaire | 12 months and 18 months
  Proportion of participants on SpoonfulONE compared to proportion of participants on the non-intervention arm who tolerated each individual food groups of the 9 selected food groups, measured through a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States